CLINICAL TRIAL: NCT01088971
Title: Effect of Duolac 7S Administration on Improving Symptom in Irritable Bowel Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cell Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CellBiotech
Record Dates: First submitted 2010-03-07; First posted 2010-03-18 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Starch

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Duolac 7S (Active Comparator)
  Interventions: Dietary Supplement: Duolac7S
- starch capsule (Placebo Comparator)
  Interventions: Dietary Supplement: starch

INTERVENTIONS:
Dietary Supplement: Duolac7S — 1 capsule two times everyday for 6 weeks
  Arms: Duolac 7S
Dietary Supplement: starch — 1capsule two times everyday for 6 weeks
  Arms: starch capsule

SUMMARY:
Gut microflora-mucosal interactions may be involved in the pathogenesis of irritable bowel syndrome (IBS). The purpose of this study is to investigate the efficacy of Duolac7S in changing the colonic microflora and improve the symptoms in IBS sufferers. In all, 64 patients with Rome III positive diarrhea type IBS will complete a 6-week multiple centre controlled clinical trial. Patients will be randomized to receive either 2 capsules/day Duolac7S or 2 capsules/day placebo. IBS symptoms will be monitored and scored according to Likert scale. Changes in faecal microflora, stool frequency and form, quality of life (QOL) scores will be also monitored.

ELIGIBILITY:
Inclusion Criteria:

* age: 18~65 years
* diarrhea type irritable bowel syndrome (by ROME III criteria)
* no organic bowel disease (by colonoscopy or barium enema)

Exclusion Criteria:

* pregnant women or nursing mothers
* hypersensitivity to probiotics
* congestive heart failure or ischemic heart disease
* systolic blood pressure : more than 160 mmHg or diastolic blood pressure: more than 100 mmHg
* uncontrolled diabetes mellitus, secondary dyslipidemia, hyperthyroidism, or hypothyroidism
* abdominal surgery (exception: appendectomy, hernia surgery)
* more than moderate alcohol drinking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The improvement of IBS symptoms | 6 weeks (symptom diary and weekly questionnaire)
  IBS symptoms were recorded on diary cards every evening during the treatment periods. Abdominal pain, discomfort,urgency and bloating were recorded (score 0-10); stool frequency as number of stools per day; stool consistency according to Bristol stool scale form (score 1-7).

SECONDARY OUTCOMES:
Changes in fecal microflora | baseline and after 6weeks
Changes of biochemical marker | baseline and after 6weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Gangnam Severance Hospital, Seoul, Seoul, South Korea